CLINICAL TRIAL: NCT06550570
Title: Evaluation of the Impact of Ambulatory Epidural on Maternal Satisfaction During Delivery and Postpartum
Acronym: PERIDEAMBU
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02Obs-CHRMT
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-08

CONDITIONS: Childbirth; Epidural; Anesthesia
Keywords: Maternal satisfaction; ambulatory epidural; physiology; analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional epidural anesthesia (=before revision of the usual practice of the maternity ward): A local anesthetic and an opioid are administered into the epidural space, as per department protocol (usual practice).
  Interventions: Behavioral: QEVA questionnaire
- Ambulatory epidural anesthesia (=after revision of the usual practice of the maternity ward): Low doses of local anesthetic and an opioid are administered into the epidural space to allow the patient to walk around while being monitored, as per department revised protocol (usual practice)
  Interventions: Behavioral: QEVA questionnaire

INTERVENTIONS:
Behavioral: QEVA questionnaire — QEVA questionnaire administered at 2 days pospartum (in hospital) and 4 weeks postpartum (phone call). (specific for the study)

SUMMARY:
Childbirth is a special event for women. Maternal satisfaction regarding childbirth is quite important, that is why this factor has to be taken into account. A bad experience related to childbirth could lead to serious psychological and organic consequences such as postpartum depression, mother-baby bond deterioration and chronic pelvic pain. Childbirth image changed over the years to the extent that an increasingly physiological process keeping analgesia and safety is more and more desired. In this perspective, this study aims to investigate an approach so-called ambulatory epidural. Indeed, only a few studies have been conducted and the ones published in 1990s did not involve the current recommended pharmacological protocols.

DETAILED DESCRIPTION:
This is a multi-centre prospective observational analytical before/after-type study.

Practice changes are planned in concerned departments, in particular regarding usual patient care. This observational study aims to quantify the impact of practice changes on patient experience using a Childbirth Assessment Questionnaire (QEVA). During the "before" period, patients will receive a conventional epidural while the others, during the "after" period, will receive an ambulatory epidural. The women involved into this study must fill the QEVA form 2 days after giving birth (at the maternity) then 4 weeks after giving birth in order to get a feedback related to postpartum feelings (phone call).

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years old
* with Physiological pregnancy (fetus cephalic position, normal fetal heart rate, spontaneous work between 37 and 41 SA)
* Having benefited from epidural, usual or ambulatory depending on the study period
* who speeks and understand French
* who signed a free and informed consent form

Exclusion Criteria:

* Hearing or comprehension impairment
* Twin pregnancies
* Scarred uterus
* Fetus in non cephalic position
* Imminent delivery
* Women under protective supervision (guardianship, curatorship)
* Women bereaved of a spouse or child during pregnancy
* Hospitalization of child in neonatology after delivery
* Women hospitalized in critical care units after childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Birthgiving women
Study Population: Pregnant women willing to give birth at CHR Metz/Thionville (maternity)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-07-23 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
Obstetrical labor and delivery experience in birthgiving women | at 2 days postpartum
  The "emotional state" dimension of the Childbirth Assessment Questionnaire (QEVA) will be evaluated.
  This questionnaire is written and validated in French. It contains 26 questions covering 4 dimensions: emotional state, relations with nursing staff, first moments with the baby, and the young mother's feelings one month before delivery.

SECONDARY OUTCOMES:
Relations with nursing staff and first moments with the child | at 2 days postpartum
  Other dimensions and isolated items of the QEVA questionnaire
Obstetrical labor and delivery experience in birthgiving women | at 4 weeks postpartum
  " emotional state " dimension of the Childbirth Assessment Questionnaire (QEVA)
Labor and delivery safety : time spent in the delivery room | at 2 days postpartum
  Time spent in the delivery room (min)
Labor and delivery safety: need for instrumental extraction | at 2 days postpartum
  Need for instrumental extraction (yes/no)
Labor and delivery safety : emergency caesarean sections | at 2 days postpartum
  Emergency caesarean sections (yes/no),
Labor and delivery safety: ability to maintain spontaneous micturition | at 2 days postpartum
  Ability to maintain spontaneous micturition (yes/no)
Safety of ambulation | at 2 days postpartum
  absence of the following events : motor block, hypotension, malaise, falls, difficulty in achieving ambulation

CONTACTS AND LOCATIONS:
Overall Officials: Lisa LEON, MD, Principal Investigator — CHR Metz Thionville Hopital Femme Mère Enfant
Locations (2):
- France (2):
  - CHR Metz Thionville Hopital Femme Mère Enfant, Metz
  - CHR Metz-Thionville Hopital Mère Enfant, Thionville

IPD SHARING:
Plan to Share IPD: No